CLINICAL TRIAL: NCT06632808
Title: Effects of Deep Cervical Flexor Muscle Exercises on Pain, Spinal Posture, and Sensory Sensitivity in Patients With Tension-Type Headache: A Single-Blind Randomized Controlled Trial
Brief Title: Effectiveness of Deep Cervical Flexor Muscle Exercises in Patients With Tension-Type Headache
Acronym: Single-Blind
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Tension-Type Headache
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-07

CONDITIONS: Tension-Type Headache
Keywords: Tension-type headache; Pain; Posture; sensory sensitivity
MeSH Terms: conditions — Tension-Type Headache; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep cervical flexor muscle exercises (Experimental): deep cervical flexor muscle exercises program
  Interventions: Other: Exercise
- Control (No Intervention): no intervention

INTERVENTIONS:
Other: Exercise — Deep cervical flexor muscle exercises target the deep neck muscles that play a crucial role in the stabilization of the cervical spine and the maintenance of proper posture. These muscles, particularly the longus colli and longus capitis, are responsible for the correct alignment of the head and neck. The exercises typically involve gentle flexion of the neck (bringing the chin towards the chest) with low-intensity, controlled movements. The goal is to strengthen these muscles, enhance spinal stability, and alleviate symptoms such as tension-type headaches. Additionally, these exercises support postural control and can reduce excessive strain on the neck.
  Arms: deep cervical flexor muscle exercises

SUMMARY:
The aim of this study is to evaluate the effects of deep cervical flexor muscle exercises on pain, spinal posture, and sensory sensitivity in patients with tension-type headaches. Designed as a single-blind randomized controlled trial, the study will assess participants' pain levels using the Visual Analog Scale (VAS), sensory sensitivity through the Sensory Sensitivity Scale, and spinal posture via a digital inclinometer for objective measurements. This research seeks to determine the effectiveness of these exercises in managing pain, improving spinal posture, and contributing to the enhancement of sensory sensitivity.

DETAILED DESCRIPTION:
The objective of this study is to comprehensively evaluate the impact of deep cervical flexor muscle exercises on three key outcomes in patients suffering from tension-type headaches: pain intensity, spinal posture, and sensory sensitivity. Tension-type headaches, often associated with poor posture and muscular dysfunction, can significantly affect daily functioning and quality of life. This study seeks to explore whether targeted exercises for the deep cervical flexor muscles can alleviate these symptoms.

Designed as a single-blind randomized controlled trial, this research will involve carefully selected participants who will be randomly assigned to either an intervention group or a control group. The intervention group will undergo a structured exercise regimen focusing on deep cervical flexor muscles, while the control group will not receive this specific intervention.

To measure the effectiveness of the intervention, three primary assessment tools will be employed: pain levels will be evaluated using the Visual Analog Scale (VAS), which provides a subjective yet widely accepted measure of pain intensity; sensory sensitivity will be assessed using the Sensory Sensitivity Scale, offering insight into changes in sensory perceptions related to the headache condition; and spinal posture will be objectively measured using a digital inclinometer, which quantifies postural alignment and deviations.

This research aims to contribute to the understanding of non-pharmacological interventions for tension-type headaches, providing evidence on whether deep cervical flexor exercises can reduce pain, improve spinal posture, and positively influence sensory sensitivity, potentially offering a holistic approach to managing these chronic headaches.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with tension-type headache

Exclusion Criteria:

* whiplash injury,
* significant neck trauma (caused by trauma to the neck, fracture, distortion, or violent attack that have caused the current NP),
* nerve root compression of the cervical spine,
* persistent headache attributed to traumatic injury to the head
* cluster headache,
* trigeminal neuralgia,
* pregnancy,
* breastfeeding,
* severe physical and/or mental illness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2025-01-24 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Two months
  VAS is used to convert some values that cannot be measured numerically into numerical values. Two extreme definitions of the severity of pain are written on both ends of a 10 cm line and the patient is asked to indicate his/her own condition by placing an X mark on the line where he/she deems appropriate.
Sensory Sensitivity Scale | Two months
  Sensory Sensitivity Scale: is a tool used to diagnose sensory modulation problems clinically. The Sensory Sensitivity Scale has two parts; the first part asks the person to relate to the intensity of the responses, while the second part asks the person to relate to the frequency of the responses. The scale consists of sensory stimuli including auditory, visual, taste, smell, vestibular (kinesthesia) and somatosensory (proprioceptive and tactile) stimuli except pain.